CLINICAL TRIAL: NCT01418872
Title: A Cluster-Randomized Clinical Trial Of Two Educational Strategies In Cardiovascular Health (CVH) In Child Population. The Savinghearts Project
Brief Title: A Clinical Trial Of Two Educational Strategies In Cardiovascular Health In Child Population
Acronym: SAVINHEARTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Agencia Lain Entralgo (Other Government)
Collaborators: Gerencia de Atención Primaria, Madrid (Other Government); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Instituto de Salud Carlos III (Other Government); Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Comunidad de Madrid (Other)
Responsible Party: Principal Investigator, Blanca Novella, Médico familia SERMAS, Agencia Lain Entralgo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1668-BK-148
Record Dates: First submitted 2011-08-12; First posted 2011-08-17 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Obesity; Cardiovascular Diseases Prevention; Paediatrics
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Breakfast (Active Comparator): The activity will be performed at the school dining hall, scheduling 1 hour for breakfast,within the school hours, with maximum 50 children per turn It involves placing a table mat, a cup, a plate and two slices of bread per child, plus 1-liter bottle of milk for each four children and 1-liter bottle of oil for each twelve. The dining hall will be all set up before the students come in.
  Participatory lesson : Ideal number of daily meals, Importance of daily breakfast for the activity, Time for breakfast, Basic components for a healthy breakfast, The role of cereals at breakfast, The role of dairy products at breakfast,The role of fruits at breakfast, Importance of exercise for cardiovascular health, The role of unhealthy habits: sedentary lifestyle.
  The students will be invited to take the table mat and the cup, in which is inscribed: "I am a heart-saver", so that they take them home and serve as a reminder of the activity.
  A pamphlet of the NAOS strategy will also be delivered.
  Interventions: Other: Didactic Concerts
- Didactic concerts (Experimental): The activity we are going to test consists in a communication and spreading strategy.
  The activity will take place in the auditorium of the school, scheduling 1 hour for concert, within the school hours, and having maximum 50 children per turn.
  Preparation of the auditorium for the activity 5 classic musical pieces and a story as a conducting thread. Children will be asked to clap and raise hands to participate in the mission of becoming a heart-savers: Ideal number of daily meals, Importance of daily breakfast for the activity, Time for breakfast, Basic components for a healthy breakfast, The role of cereals at breakfast, dairy products in breakfast, fruits at breakfast, Importance of exercise for cardiovascular health, The role of sedentary lifestyle.
  Students will be invited to take the playbill as a bookmark format and a cup is inscribed: "I am a heart-saver", so that they take them home and serve as a reminder of the activity. A NAOS strategy pamphlet will also be delivered.
  Interventions: Other: Didactic Concerts

INTERVENTIONS:
Other: Didactic Concerts — The activity we are going to test consists in a communication and spreading strategy.
  The activity will take place in the auditorium of the school, scheduling 1 hour for concert, within the school hours, and having maximum 50 children per turn.
  Preparation of the auditorium for the activity 5 classic musical pieces and a story as a conducting thread. Children will be asked to clap and raise hands to participate in the mission of becoming a heart-savers: Ideal number of daily meals, Importance of daily breakfast for the activity, Time for breakfast, Basic components for a healthy breakfast, The role of cereals at breakfast, dairy products in breakfast, fruits at breakfast, Importance of exercise for cardiovascular health, The role of sedentary lifestyle.
  Students will be invited to take the playbill as a bookmark format and a cup is inscribed: "I am a heart-saver", so that they take them home and serve as a reminder of the activity. A NAOS strategy pamphlet will also be delivered.

SUMMARY:
AIM: To evaluate the effectiveness of two strategies in cardiovascular risk in children 2º grade in the community of Madrid.

DESIGN: cluster-randomized trial with blinded evaluator SCOPE AND SUBJECTS OF STUDY: Children of both sexes enrolled in 2º grade in public schools in the community of Madrid. Rate exclusion criteria INTERVENTION: Schools were randomly assigned to two groups: an experimental group that the investigators organized a concert teaching focused on messages cardio, a second group or control group to which they will host a healthy breakfast as it has been offering the Community of Madrid .

MEASUREMENTS: The primary end result is the increase of correct answers on a standardized test to be administered before and after the activity.

Secondary outcomes will be, improving the same questionnaire at 6 months and reduced overall weight and center from before the intervention at 6 months of it.

ELIGIBILITY:
Inclusion Criteria:

* 2º grade of primary school students present the day of the activity, whose parents had signed the informed consent to participate in the study and with no exclusion criteria at the moment of the intervention

Exclusion Criteria:

* Students with food allergies or intolerances.
* Students with severe hearing impairment (not corrected).
* Students whose parents didn´t sign the informed consent to participate in the study.
* Students with a poor understanding of oral and written language.
* To have previously received healthy breakfasts interventions or educational concerts.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1730 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge and attitudes in Cardiovascular Health | Before the intervention (baseline) and 7 days after and 6 months after the intervention.
  The primary outcome variable will be the changes in healthy heart knowledge and attitudes in children in 2º grade of primary school. We will measure this primary outcome variable using 2 modified INUTCAM questionnaires

SECONDARY OUTCOMES:
Body Mass Index (BMI) | before the intervention (baseline) and 6 months after them.
  The secondary outcome variable will be BMI measured at the moment of the intervention and 6 months after it.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Novella, PhD, Principal Investigator — SERMAS
Locations (1):
- Agencia Lain Entralgo, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Sanchez-Gomez LM, Fernandez-Luque MJ, Ruiz-Diaz L, Sanchez-Alcalde R, Sierra-Garcia B, Mayayo-Vicente S, Ruiz-Lopez M, Loeches-Belinchon P, Lopez-Gonzalez J, Gonzalez-Gamarra A, Gallego-Arenas A, Cubillo-Serna A, Gil-Juberias G, Perez-Cayuela P, Canedo-Arguelles CA, Garcia-Pascual JN, Ruiz-Chercoles E, Suarez-Fernandez C, Garcia-Polo I, Abad-Perez D, Ballesteros-Arribas JM, Izquierdo-Martinez M, Salvador-Alcaide E, Arribas-Vela AB, Alonso-Perez JM, Veja-Piris L, Rodriguez-Salvanes F, Novella-Arribas B. A cluster-randomised clinical trial comparing two cardiovascular health education strategies in a child population: the Savinghearts project. BMC Public Health. 2012 Nov 23;12:1024. doi: 10.1186/1471-2458-12-1024. PMID 23176593